CLINICAL TRIAL: NCT01631643
Title: One Touch® Verio®IQ European Clinical Outcomes Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision to withdraw trial
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3093513
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes
Keywords: Blood glucose monitor; Pattern management; Pattern guide; Education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: One Touch VerioIQ Blood Glucose Monitor — BGM with pattern alert technology and with associated pattern guide

SUMMARY:
Evaluation of the clinical benefits of One Touch VerioIQ system.

DETAILED DESCRIPTION:
Evaluation of the clinical benefits of the One Touch VerioIQ system. The system contains pattern alert technology and comes with educational material (Pattern guide) which provides additional support and insights to patients and health care providers to help them make more informed decisions during blood glucose management.

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 18 to 80 years old
* ADA guidelines for FPG and PPG appropriate
* A1C greater or equal to 8.0% and less than or equal to 10.5%
* lab A1C greater than or equal to 8.0% in the last 6-12mths
* Diagnosed with type 1 or 2 in at least last 1 year
* on stable dose of OADs for at least 3mths prior to screening
* willingness to test 7 BGM tests per day
* willing to remain on same therapy as baseline (MDI) for duration of study

Exclusion Criteria:

* unlikely to be compliant to study procedures
* has or has currently used One Touch VerioIQ
* Is on fixed doses of insulin for MDI therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change in A1C from baseline to week 24 | 24 weeks
  A1C (also known as hemoglobin A1C or glycosylated hemoglobin)

SECONDARY OUTCOMES:
Change in A1C from baseline to week 12 | 12 weeks
Change in FPG from baseline to 24 weeks | 24 weeks
  FPG (Fasting plasma glucose)
Change in proportion of subjects with A1C less than or equal to 7.0% at week 24 | 24 weeks
Change in 30 day mean glucose comparing first month to last month after 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Thivolet, MD, Principal Investigator — Centre Hospitalier Lyon Sud